CLINICAL TRIAL: NCT03587922
Title: Post Market Study of the FANTOM Sirolimus-Eluting Bioresorbable Coronary Scaffold
Brief Title: FANTOM Post Market Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: REVA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCT6700
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Single arm study with treatment of Fantom scaffold
  Interventions: Device: Fantom

INTERVENTIONS:
Device: Fantom — Treatment of den ovo coronary lesions

SUMMARY:
Post Market study of the Fantom Sirolimus-Eluting Bioresorbable Coronary Scaffold

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age.
* The subject must have evidence of myocardial ischemia
* The patient is an acceptable candidate for PTCA, stenting and emergent CABG.
* The patient is willing and able to comply with the specified follow-up evaluations.
* The patient's written informed consent has been obtained.

Each lesion to be treated with Fantom must meet all the following baseline criteria:

* De novo lesion in a native coronary artery
* Visually estimated stenosis of > or equal to 50% and <100%.
* Visually estimated RVD > or equal to 2.5 mm and less than or equal to 3.75 mm.
* Baseline TIMI flow greater than or equal to 2 per visual estimate.
* Lesion Length less than or equal to 20 mm, able to be covered by a single scaffold
* No angiographic complications (e.g. distal embolization, side branch closure).
* No dissections greater than or equal to NHLBI type C.
* Patient has no ongoing chest pain or ECG ST-segment of T-wave changes.

Exclusion Criteria:

* The patient has a known allergy, intolerance, or is contraindicated to aspirin, both heparin and bivalirudin, clopidogrel and/or contrast media, and cannot be adequately pre-medicated.
* The patient has experienced an acute ST-segment elevation myocardial infarction (AMI: STEMI) within 72 hours of the procedure and either CK-MB or Troponin has not returned to within ULN (Note: the patient with a recent NSTEMI with elevated biomarkers may still be enrolled).
* The patient has a left ventricular ejection fraction of <30%.
* The patient has unprotected left main coronary disease with greater than or equal to 50% stenosis.
* The patient has undergone prior PCI within the target vessel during the last 12 months.
* Prior PCI of a non-target vessel within 24 hours prior to the procedure, or within 30 days prior to the procedure if unsuccessful or complicated. Note: Prior PCI of a non-target vessel is acceptable if performed anytime > 30 days before the index procedure or between a minimum of 24 hours and 30 days before the index procedure is successful and uncomplicated.
* Prior PCI within 3 years with a bioresorbable scaffold in any vessel.
* The patient requires future staged PCI of any lesion other than a target lesion identified at the time of the index procedure.
* The patient has received any solid organ transplant or is on a waiting list for any solid organ transplant.
* At the time of screening, the subject has a malignancy that is not in remission.
* The patient is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy.
* The patient has a stent located within 3 mm of the target lesion borders.
* The target vessel is totally occluded (TIMI Flow 0 to 1).
* Excessive proximal tortuosity, vessel hinging at the lesion location or lesion angulation, such that in the operator's judgment it is unlikely that the Fantom Bioresorbable Coronary Scaffold or a standard scaffold could be delivered and/or expanded.
* The patient is currently participating in another investigational drug or device trial that has not reached its primary endpoint assessment
* The patient has co-morbidities which reduce life expectancy to less than or equal to 24 months, or a condition that may interfere with the follow-up procedures of this protocol.

The patient has:

* Known hepatic impairment (liver function tests (SGOT, SGPT, or ALT) >3 times normal);
* Known impaired renal function (serum creatinine greater than or equal to 2.5 mg/dL).
* A platelet count <100,000 cells/mm3 and/or >700,000 cells/mm3
* The patient has a history of stroke (CVA) or TIA within the prior 6 months, or any permanent neurologic defect, or any prior history of intracerebral bleeding.
* The patient has an active peptic ulcer or upper GI bleeding within the prior 6 months.
* The patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* The patient is a woman that is pregnant or lactating or is planning to get pregnant during the follow-up period of this trial. Note: Women of child-bearing potential should have a negative pregnancy test before enrollment.
* Target lesion ostial (within 3mm of vessel origin).
* Target lesion is located in the left main or there is a > 30% diameter stenosis in the left main artery
* Target lesion has moderate to severe calcification.
* Target segment(s) has one or more side branches >2.0 mm in diameter.
* Target segment(s) has a side branch with either an ostial or non-ostial lesion with diameter stenosis >50% or requiring dilation
* Target lesion is located within an arterial bypass graft conduit or saphenous vein graft.
* Target lesion is located within a previously stented region.
* Target lesion is located within a segment supplied by distal graft.
* Target lesion has possible or definite thrombus.
* The patient is currently receiving or will require chronic anticoagulation therapy (e.g. coumadin, dabigatran, apixaban, rivaroxaban, or edoxaban for any reason).
* The patient is known to need or has a planned surgical procedure or any other reason is present which might require discontinuing aspirin and/or clopidogrel within 1 year of the Fantom scaffold implantation
* Patient has a known allergy to tyrosine derived polycarbonate or Sirolimus and its structurally related compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure | 12 Months
  TLF Composite defined by rate of Cardiac Death, Target Vessel MI and Ischemic Driven Target Lesion Revascularization

CONTACTS AND LOCATIONS:
Locations (10):
- Wilhelminenhospital, Vienna, Austria
- Germany (8):
  - Juedisches Krankenhaus Berlin, Berlin
  - Technische Universitat Dresden, Dresden
  - Universitatsklinikum Halle, Halle
  - Klinikum Herford, Herford
  - Universitatsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Clemenshospital Muenster, Münster
  - Klinkum Oldenburg, Oldenburg
  - Marien Hospital Witten, Witten
- University Kantonsspital Baselland, Liestal, Switzerland

IPD SHARING:
Plan to Share IPD: No